CLINICAL TRIAL: NCT04462016
Title: Blood Glucose Response to a Calamansi Drink in Healthy Adults
Brief Title: Effects of Calamansi on Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Malaysia Sarawak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MDP20505_2017/2018_MS0001
Record Dates: First submitted 2020-07-01; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Blood Glucose Response
Keywords: calamansi; glycaemic index; post-prandial blood glucose
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference drink (Active Comparator): Healthy volunteers' blood glucose response to reference drink (glucose)
  Interventions: Other: Glucose
- Test drink (Experimental): Healthy volunteers' blood glucose response to test drink (calamansi)
  Interventions: Other: Calamansi

INTERVENTIONS:
Other: Calamansi — 250 ml of a commercially sourced calamansi drink
  Arms: Test drink
Other: Glucose — 75 g of glucose dissolved in 250 ml of drinking water
  Arms: Reference drink

SUMMARY:
It is important to bring the blood glucose levels of those with type 2 diabetes mellitus (T2DM) back to normal levels as this can stop the condition from worsening and prevent other conditions that are related to T2DM from developing. One way to maintain healthy blood glucose level is the use of the glycaemic index (GI), which ranks food according to how the body responds to its carbohydrate content. Low GI foods corresponds to low increase in blood glucose levels. Calamansi is a citrus that is believed not to induce an increase in blood glucose levels. Since beverages from calamansi are available and diabetes is a health concern in the community, it is important to investigate the effect of consuming this drink. Finger prick blood were tested in order to obtain the blood glucose levels for calculating the GI for the calamansi drink.

ELIGIBILITY:
Inclusion Criteria:

* non-smoker
* BMI between 18.5 and 24.99 kg/m2
* waist circumference less than 102 cm
* random blood glucose less than 7.8 mmol/L
* negative urine dipstick result
* not on any medications
* no family history of inherited diseases
* no heart conditions (angina, arrhythmia or heart failure)
* no history of acute medical or surgical event within the past 6 months.

Exclusion Criteria:

* pre-existing conditions such as HIV, hepatitis, inflammatory bowel diseases, diabetes mellitus, kidney disease, blood disorders (such as thalassaemia)

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline blood glucose levels | 30, 60, 90, 120 min after drinking
  Capillary blood glucose using glucometer

SECONDARY OUTCOMES:
Change from baseline urinary glucose levels | 30, 60, 90, 120 min after drinking
  Dipstick test

CONTACTS AND LOCATIONS:
Overall Officials: Angela Siner, PhD, Principal Investigator — Universiti Malaysia Sarawak
Locations (1):
- Faculty of Medicine and Health Sciences, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: This will be made available starting 6 months from the date of publication; for the next 5 years.
Access Criteria: Through reasonable request to the corresponding author.

REFERENCES:
- [Derived] Siner A, Sevanesan MS, Ambomai T, Abd Wahab Z, Lasem L. Blood glucose response to a calamansi drink in healthy adults: a non-randomised study. BMC Res Notes. 2020 Aug 28;13(1):404. doi: 10.1186/s13104-020-05250-8. PMID 32859257